CLINICAL TRIAL: NCT01361594
Title: Intensive Insulin Therapy in Patients Undergoing Coronary Artery Bypass Surgery
Acronym: CABG
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Principal Investigator, Guillermo Umpierrez, Professor of Medicine, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00048356; 00048356-2010 (Other: Other)
Record Dates: First submitted 2011-02-03; First posted 2011-05-27 (Estimated); Results first posted 2014-12-31 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-12

CONDITIONS: Diabetes
Keywords: Diabetes; Coronary Artery Bypass Surgery; Glycemic control; Insulin infusion
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intensive insulin treatment (Active Comparator): Intensive insulin treatment (BG target: 100-140 mg/dL)
  Interventions: Other: Regular insulin (intensive treatment)
- Conventional insulin treatment (Active Comparator): Conventional insulin treatment (BG target: 141-180 mg/dl)
  Interventions: Other: Regular Insulin (conventional treatment)

INTERVENTIONS:
Other: Regular insulin (intensive treatment) — Titration of the IV insulin rate for glucose goal 100-140 mg/dL
  Arms: Intensive insulin treatment
Other: Regular Insulin (conventional treatment) — Titration of the IV insulin rate for glucose goal 141-180 mg/dl
  Arms: Conventional insulin treatment

SUMMARY:
High blood glucose levels (hyperglycemia) in cardiac surgery patients with diabetes are associated with increased risk of hospital complications. Blood sugar control with intravenous insulin may prevent such hospital complications. Many patients undergoing cardiac bypass surgery (CABG) develop high blood sugars and require insulin therapy (shortly before or after surgery). It is not clear what the best insulin regimen is or what is the best blood sugar target in these patients. Accordingly, this research study aims to determine optimal blood glucose levels during the in patients undergoing cardiac bypass surgery. Patients will be divided in two groups. The intensive insulin group will be maintained at blood glucose between 100-140 mg/dl and the conventional treatment group at a glucose level between 140-180 mg/dl. The insulins to be used in this trial (lantus, aspart and regular insulin) are approved for use in the treatment of patients with diabetes by the FDA (Food and Drug Administration). A total of 326 patients with high blood glucose after cardiac bypass surgery will be recruited in this study. Patients will be recruited at Emory University Hospital, Emory Midtown Hospital and Grady Memorial Hospital.

DETAILED DESCRIPTION:
Several prospective cohort studies as well as randomized clinical trials (RCT) in cardiac surgery patients have shown that intensified insulin therapy (target BG: 110-140 mg/dl) results in a reduction in short- and long-term mortality compared with conventionally treated patients. The results of recent international trials in critically ill patients; however, have failed to show a significant improvement in mortality or have even shown increased mortality risk as well as increased number of hypoglycemic events with intensive compared to less intensive glycemic control. Based on the results of these ICU trials, new ADA and AACE guidelines recommended a glycemic target between 140 and 180 mg/dl in the ICU including cardiac surgery patients. There is concern that such high BG targets might increase the risk of hospital complications in cardiac surgical patients in whom intensive glucose control has consistently reduced infections, length of hospital stay, resource utilization, and cardiac-related mortality. The overall objective of this proposal is to conduct the first prospective RCT to determine the optimal BG target during the perioperative period in hyperglycemic subjects who undergo CABG in the United States. Subjects will be randomized to undergo intensive insulin therapy adjusted to maintain a BG between 100 mg/dl and 140 mg/dl or to a conventional glucose control with a target BG between 141 mg/dl and 200 mg/dl in the ICU. The central hypothesis of this proposal is that intensive insulin management will reduce perioperative complications compared to a conventional BG control in cardiac surgery patients.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females between the ages of 18 and 80 years undergoing CABG +/- valve surgery.
2. Post surgical hyperglycemia (BG > 140 mg/dl).
3. Patients with and without a history of type 2 diabetes

Exclusion Criteria:

1. Patients requiring combination CABG with additional procedures such aorta replacement.
2. Patients with severely impaired renal function (serum creatinine ≥3.0 mg/dl or GFR < 30 ml/min) or clinically significant hepatic failure.
3. Subjects with acute hyperglycemic crises such as diabetic ketoacidosis (DKA) and hyperosmolar hyperglycemic state.
4. Moribund patients and those at imminent risk of death (brain death or cardiac standstill).
5. Patients or next-to-kin with mental condition rendering the subject or family member unable to understand the nature, scope, and possible consequences of the study.
6. Female subjects who are pregnant or breast-feeding at time of enrollment into the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 338 (Actual)
Dates: Start 2011-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo E Umpierrez, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Emory University Hospital, Emory University Hospital - Midtown and Grady Hospital
Pre-assignment Details: Patients undergoing coronary artery bypass surgery (CABG) that develop hyperglycemia (defined as a blood glucose >140) intraoperatively or in an intenstive care unit (ICU) post-surgical procedure. 33 patients withdrawn prior to randomization, due to various reasons, including surgery cancellation, transportation to a different hospital, etc.
Period: Overall Study
Arm/Group | Intensive Insulin Treatment | Conventional Insulin Treatment
Started | 152 | 153
Completed | 151 | 151
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Population: Only subjects that completed the study were accounted for in the baseline characteristics.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intensive Insulin Treatment | Conventional Insulin Treatment | Total
Number analyzed (Participants) | 151 | 151 | 302
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 79 | 80 | 159
  >=65 years | 72 | 71 | 143
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 39 | 84
  Male | 106 | 112 | 218

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects That Were Diagnosed for Peri-operative Complications
Description: Number of participants that presented at least 1 complications including sternal wound infection, bacteremia, acute renal failure, respiratory failure, and major cardiovascular events (MACE) during the current hospitalization and up to 6 months after hospitalization
Time Frame: Within 6 months of hospitalization
Measure: Number; unit: participants
Arm/Group | Intensive Insulin Treatment | Conventional Insulin Treatment
Number analyzed (Participants) | 151 | 151
participants | 58 | 70

2. Secondary Outcome: Glycemic Control
Description: 1. Hyperglycemic events (BG > 200 mg/dL) in ICU and non-ICU
  2. Hypoglycemic events (BG < 70 mg/dl; severe hypoglycemia (BG < 40 mg/dl).
Time Frame: average 1 month during the hospitalization
Reporting Status: Not Posted

3. Secondary Outcome: Major Cardiovascular Events
Description: 1. Acute myocardial infarction : (1) typical increase and gradual decrease (troponin) or (2) more rapid increase and decrease (creatine kinase MB) of biochemical markers of myocardial necrosis with at least one of the following: (a) ischemic symptoms, (b) development of pathologic Q waves on the electrocardiogram, (c) electrocardiographic changes indicative of ischemia (ST-segment elevation or depression), or (d) coronary artery intervention (e.g., coronary angioplasty).
  2. Congestive heart failure
  3. Cardiac arrhythmias: malignant arrhythmia
Time Frame: average 1 month during the hospitalization
Reporting Status: Not Posted

4. Secondary Outcome: Acute Renal Failure
Description: new-onset abnormal renal function: serum creatinine > 2.0 mg/dL or an increment level > 50% from baseline
Time Frame: average 1 month during the hospitalization
Reporting Status: Not Posted

5. Secondary Outcome: Respiratory Failure, Defined as PaO2 Value < 60 mm Hg While Breathing Air or a PaCO2 > 50 mm Hg.
Description: Respiratory failure, defined as PaO2 value < 60 mm Hg while breathing air or a PaCO2 > 50 mm Hg.
Time Frame: average 1 month during the hospitalization
Reporting Status: Not Posted

6. Secondary Outcome: ICU and Hospital Length of Stay, and ICU Readmissions
Description: ICU and hospital length of stay, and ICU readmissions
Time Frame: average 1 month during the hospitalization
Reporting Status: Not Posted

7. Secondary Outcome: Surgical Wound Infection
Description: superficial and deep sternal wound infection
Time Frame: average 1 month during the hospitalization
Reporting Status: Not Posted

8. Secondary Outcome: Pneumonia (CDC Criteria)
Description: Pneumonia (CDC criteria)
Time Frame: average 1 month during the hospitalization
Reporting Status: Not Posted

9. Secondary Outcome: Cerebrovascular Events
Description: permanent stroke and reversible ischemic neurologic deficit.
Time Frame: average 1 month during the hospitalization
Reporting Status: Not Posted

10. Primary Outcome: Hospital Mortality
Description: Mortality is defined as death occurring during admission, either during ICU or after transition to non-ICU admission.
Time Frame: average 1 month during the hospitalization
Measure: Number; unit: participants
Arm/Group | Intensive Insulin Treatment | Conventional Insulin Treatment
Number analyzed (Participants) | 151 | 151
participants | 5 | 2

11. Secondary Outcome: Duration of Ventilatory Support and ICU Readmission
Description: Duration of ventilatory support and ICU readmission
Time Frame: average 1 month during the hospitalization
Reporting Status: Not Posted

12. Secondary Outcome: Thirty Day Mortality
Description: Thirty day mortality
Time Frame: within 30 days of discharge
Reporting Status: Not Posted

13. Secondary Outcome: Number of Hospital Readmissions and Emergency Room Visits
Description: Number of hospital readmissions and emergency room visits
Time Frame: Within 30 days after discharge
Reporting Status: Not Posted

14. Secondary Outcome: Incidence of Organ Failures Assessed by the Daily SOFA Score
Description: Incidence of organ failures assessed by the daily SOFA score
Time Frame: average 1 month during the hospitalization
Reporting Status: Not Posted

15. Secondary Outcome: Measures of Inflammation
Description: Measures of inflammation (C-reactive protein, TNF-alpha; IL-6) and oxidative stress markers
Time Frame: average 1 month during the hospitalization
Reporting Status: Not Posted

16. Secondary Outcome: Major Cardiovascular Events
Description: as for outcome 3
Time Frame: within 3 months after discharge
Reporting Status: Not Posted

17. Secondary Outcome: Surgical Wound Infection
Description: Superficial and deep sternal wound infection
Time Frame: within 3 months after discharge
Reporting Status: Not Posted

18. Secondary Outcome: Pneumonia (CDC Criteria)
Description: Pneumonia (CDC criteria)
Time Frame: Within 3 months after discharge
Reporting Status: Not Posted

19. Secondary Outcome: Cerebrovascular Events
Description: permanent stroke and reversible ischemic neurologic deficit
Time Frame: within 3 months after discharge
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: 3 subjects that were randomized (but no intervention started) so they were not considered to be at-risk participants for adverse events.
Arm/Group | Intensive Insulin Treatment | Conventional Insulin Treatment
Serious Adverse Events (participants affected / at risk) | 63/151 | 78/151
Other Adverse Events (participants affected / at risk) | 56/151 | 50/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intensive Insulin Treatment (N=151) | Conventional Insulin Treatment (N=151)
Acute renal failure (Renal and urinary disorders) | 21 (21) | 28 (28)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 17 (17) | 29 (29) — Intubation > 2 days
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 8 (8)
Major Adverse Cardiac Events (MACE) (Cardiac disorders) | 51 (51) | 63 (63) — defined as death, myocardial infarction, or clinically-driven target lesion revascularizations
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intensive Insulin Treatment (N=151) | Conventional Insulin Treatment (N=151)
Surgical re-intervention (Cardiac disorders) | 7 (7) | 9 (9)
ICU Re-admission (Injury, poisoning and procedural complications) | 7 (7) | 8 (8)
Hypoglycemia (ICU) (Endocrine disorders) | 12 (12) | 3 (3) — blood glucose less than 70 mg/dL but greater than 40 mg/dL
Hypoglycemia (immediately after treatment) (Endocrine disorders) | 30 (30) | 30 (30) — blood glucose less than 70 mg/dL but greater than 40 mg/dL

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes